CLINICAL TRIAL: NCT06399133
Title: Care Package for Postoperative Constipation
Acronym: Car_Package
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubra KAYA (Other)
Responsible Party: Sponsor-Investigator, Kubra KAYA, Principal Investigator, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: kübra_1
Record Dates: First submitted 2024-04-27; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Care; Constipation
Keywords: Constipation Risk; Constipation Severity; Nursing; Care; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: This was a single-center, randomized controlled trial of patients hospitalized in the Orthopedics and Traumatology Clinic of a state hospital between September 15, 2022, and April 30, 2023. Overall, 102 patients were randomly assigned to study and control groups. Routine clinical practice was maintained for patients in the control group, whereas a care package constituting postoperative warm water intake, abdominal massage, and a high-fiber diet was provided to those in the study group. Data was collected using the 'Constipation Risk Assessment Scale' and 'Visual Analog Scale'. Constipation severity was evaluated by administering the scales one day before surgery (T0) and one (T1), two (T2), three (T3), and four (T4) days postoperatively. Data were analyzed using SPSS software (version 20.0; IBM, Canada). Statistical significance was set at p < 0.05.
Masking Description: This was a single-center, randomized controlled trial of patients hospitalized in the Orthopedics and Traumatology Clinic of a state hospital between September 15, 2022, and April 30, 2023. Overall, 102 patients were randomly assigned to study and control groups. Routine clinical practice was maintained for patients in the control group, whereas a care package constituting postoperative warm water intake, abdominal massage, and a high-fiber diet was provided to those in the study group. Data was collected using the 'Constipation Risk Assessment Scale' and 'Visual Analog Scale'. Constipation severity was evaluated by administering the scales one day before surgery (T0) and one (T1), two (T2), three (T3), and four (T4) days postoperatively. Data were analyzed using SPSS software (version 20.0; IBM, Canada). Statistical significance was set at p < 0.05.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in the CG received routine postoperative clinical interventions.
- Study Group (Experimental): Patients in the SG received a care package including warm water intake, abdominal massage, and a high-fiber diet.
  Interventions: Other: Warm water intake; Other: High-fiber diet; Other: Abdominal massage

INTERVENTIONS:
Other: Warm water intake — Nurses assessed the patients' gag and swallow reflexes in the SG. Patients who experienced nausea after reflex assessment were considered to have positive reflexes and were administered warm water. Packaged water was boiled in a kettle and poured into 200 mL disposable cups. After cooling the water to 38-40°C using a thermometer, patients were instructed to drink it within 3 min.
  Arms: Study Group
Other: High-fiber diet — After initiating oral intake, the patients collaborated with a dietitian to incorporate high-fiber foods containing 30 g of fiber daily into their meal menus.
  Arms: Study Group
Other: Abdominal massage — Patients in the SG received abdominal massages twice a day, in the morning from 08:00 to 09:00 and in the evening from 19:00 to 20:00, for 15 min per session, starting one day postoperatively.
  Arms: Study Group

SUMMARY:
Background: Postoperative constipation is a common complication. The effectiveness of a care package constituting warm water intake, abdominal massage, and a high-fiber diet has not been investigated in patients undergoing orthopedic surgery.

Aim: the investigators determined the effects of a care package, including warm water intake, abdominal massage, and high-fiber diet, on constipation prevention, aiming to improve patient quality of life during the postoperative period and support nurses in clinical practice.

Study design: This was a single-center, randomized controlled trial of patients hospitalized in the Orthopedics and Traumatology Clinic of a state hospital between September 15, 2022, and April 30, 2023. Overall, 102 patients were randomly assigned to study and control groups. Routine clinical practice was maintained for patients in the control group, whereas a care package constituting postoperative warm water intake, abdominal massage, and a high-fiber diet was provided to those in the study group. Data was collected using the 'Constipation Risk Assessment Scale' and 'Visual Analog Scale'. Constipation severity was evaluated by administering the scales one day before surgery (T0) and one (T1), two (T2), three (T3), and four (T4) days postoperatively. Data were analyzed using SPSS software (version 20.0; IBM, Canada). Statistical significance was set at p < 0.05.

DETAILED DESCRIPTION:
INTRODUCTİON Constipation is a common complication observed in patients undergoing orthopedic surgery. The incidence of constipation is reported to be between 40-72% in these patients . Factors such as immobilization during the postoperative period, opioid use, addressing voiding and bowel movements in bed, pain, and inadequate intake of food and fluids contribute to increased susceptibility to constipation in patients undergoing orthopedic surgery. Prolonged immobilization of patients undergoing orthopedic surgery and the widespread use of opioid analgesics in pain management protocols can increase the frequency of constipation. Additionally, increased catecholamine release due to surgical stress is considered a cause for decreased bowel mobility, leading to constipation during the postoperative period.

Constipation can lead to multiple adverse effects in patients, such as discomfort, bloating, pain, loss of appetite, nausea, vomiting, and increased psychosocial stress. Prevention and reduction of constipation symptoms improve patient comfort and quality of life. Constipation in surgical patients increases the risk of postoperative complications and prolongs hospital stay .

Multiple studies have utilized non-pharmacological methods to prevent constipation. The effects of abdominal massage and a high-fiber diet were investigated in studies aimed at preventing constipation in patients undergoing orthopedic surgery. However, no study has investigated the effects of early warm water intake on constipation in patients undergoing orthopedic surgery. Nevertheless, one study found that patients administered warm water postoperatively experienced earlier bowel movements.

The benefits of implementing care packages have been reported; however, the literature on care packages aimed specifically at preventing constipation remains limited. Several existing care packages have been reported to be effective in preventing constipation . However, no study investigated the effects of a triple care package constituting early postoperative warm water intake, abdominal massage, and a high-fiber diet on constipation prevention in patients undergoing orthopedic surgery, and previous studies have focused on individual components of the investigated care package.

AIMS AND HYPOTHESİS We aimed to determine the effects of a three-intervention constipation prevention care package constituting early postoperative warm water intake, abdominal massage, and a high-fiber diet on the severity of postoperative constipation in patients undergoing orthopedic surgery. We aimed to improve patients' quality of life and to support nurses in clinical practice during the postoperative period. Our study contributes to the literature owing to the lack of studies that investigated the effects of the aforementioned care package on constipation prevention in patients undergoing orthopedic surgery.

The following hypotheses were tested in this study:

H11: The constipation prevention care package shortens the time to first defecation postoperatively in patients undergoing orthopedic surgery.

H12: The constipation prevention care package reduces postoperative constipation severity in patients undergoing orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years,
* undergoing elective orthopedic surgery,
* able to read and write in Turkish,
* without any psychiatric illness or reception of psychiatric medications
* without chronic constipation or reception of constipation medications
* without abdominal wounds
* mobilization in the preoperative period
* without bandages or wraps on the arm and hand that would hinder answering questions
* ASA score <III,
* willing to participate in the study.

Exclusion Criteria:

* patients
* immobilized for ≥ 2 days postoperatively,
* with ileus within the first three days postoperatively,
* discharged or transferred to another service before three days postoperatively,
* unable to tolerate oral intake due to reasons such as a nasogastric tube or trauma-related jaw and mouth injuries in the postoperative period,
* who voluntarily withdrew from the study at any stage after volunteering to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Demographic Characteristics Form: | up to 4 weeks
  The first section included questions about the patient's sex, marital status, date of birth, education level, presence of a companion, employment status, presence of chronic diseases, use of continuous medications, type of surgery, general dietary habits, place of residence, bowel habits before surgery, and regular exercise habits. This form was administered to the patients one day before surgery.
Part 2: Constipation Risk Assessment Scale | up to 4 weeks
  This scale, developed by Richmond and Wright, has been tested for reliability and validity in Turkish by Koca et al. (2011) [18,19]. The original version of the scale had a Cronbach's alpha value of 0.50; however, it was determined to be 0.43 in the Turkish version [18,19]. Written permission to use the scale was obtained from Koca Kutlu et al. The scale constituted four sections, and scores were assigned at the end of each section. The total score was the sum of the section scores. The score range was 0-63, with higher scores indicating a higher risk of constipation[18]. Individuals scoring ≤10 were classified into the low-risk group, those scoring 11-15 into the moderate-risk group, and those scoring ≥ 16 into the high-risk group. This form was administered to the patients one day before surgery.
Part 3: Visual Analog Scale (VAS): | up to 4 weeks
  ): The VAS was first used by Pamuk et al. (2003) to determine symptoms related to constipation [20]. Symptoms such as straining, incomplete bowel emptying, constipation, pressure sensation in the rectum, severity of gas formation, and pain in the rectum were measured using the VAS. Low scores indicated mild symptoms, whereas high scores indicated severe symptoms. The VAS was administered to patients one day before surgery (T0) and one (T1), two (T2), three (T3), and four (T4) days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra KAYA, PhD, Study Director — kubra.kaya@hku.edu.tr
Locations (1):
- Orthopedics and Traumatology Clinic of Abdulkadir Yüksel State Hospital in Gaziantep., Gaziantep, Central, Turkey (Türkiye)